CLINICAL TRIAL: NCT06119737
Title: Effects of Exercise on Thyroid Stimulating Hormone Among Class-I Obese Patients With Diabetes Mellitus and Lipid Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Batool Hassan, Assistant Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Batool_H
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Intensity Continuous Training (Experimental)
  Interventions: Other: Exercise
- Resistance Training (Active Comparator)
  Interventions: Other: Exercise
- High-Intensity Interval Training (Active Comparator)
  Interventions: Other: Exercise
- 1/2- High-Intensity Interval Training (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Effects of exercises on TSH levels

SUMMARY:
Obesity is characterized by an excessive accumulation of body fat that gives rise to significant comorbidities, such as diabetes, hypertension, dyslipidemia, cardiovascular disease, and many cancers. According to WHO, Obesity is a worldwide epidemic, with an estimated 57.8% of adults worldwide expected to be classified as obese by 2030. Therefore, obesity is invariably referred to as a crucial public health problem that requires urgent attention to prevent obesity-related health outcomes. Thyroid dysfunction is often accompanied by changes in body weight and body composition, leading to obesity.

The rising risk of obesity has created susceptibility for every individual irrespective of age, gender and demography. Hence, the focus of researchers is now shifting to devising preventive strategies from the treatment approaches for obesity. To guide healthcare professionals in treating obesity, several guidelines from The Obesity Society (TOS) have been prepared that outline multiple therapies like lifestyle modifications, increased physical activities, dietary modifications, use of medications and in some cases, even surgeries are recommended. However, poor receptivity of exercise among the general population required healthcare professionals to design an exercise program that could be cost and time-effective for the patient. Hence, the present study aims to determine the effect of exercise and the documentation of the best possible exercise regime that could increase TSH among the class I obese population.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. The participants were recruited via the envelop method of simple random sampling technique into four groups: Moderate Intensity Continuous Training (MICT), Resistance Training (RT), High-Intensity Interval Training (HIIT) and ½ HIIT.

The training was based on a warm-up session of 5 to 10 minutes followed by conditioning and a cool-down phase of 5 to 10 minutes. The detailed description of each phase is as follows:

Warmup Warm-up exercises, including High Knee and Jumping Jack Exercises, were performed 5 to 10 minutes using the Lindstrom protocol to increase core body temperature and improve blood.

Conditioning Conditioning includes exercises that were performed by the participants under the supervision of a Qualified senior Physical Therapist for varied duration of time depending on the protocol of training.

Moderate Intensity Continuous Training Moderate-intensity endurance exercises were performed by the participants under the supervision of a Qualified senior Physical Therapist by using either a treadmill or cycle ergometer. Exercise frequency was 3 days per week for 16 weeks, each session lasting for 30 minutes. The intensity was calculated using the Karovonean method10, in which a targeted heart rate of 60-85% was maintained for the purpose of conditioning.

THR= (MHR-RHR x Training %) + RHR

Resistance Exercise Conditioning using resistance exercises involves training of 11 major muscle groups of the body that include i) biceps, ii) triceps, iii) deltoid, iv) trapezius, v) latisimus dorsi, vi) pectoralis major vii) abdominals, viii) back extensors, ix) hamstrings, x) quadriceps, and xi) calf (WLC). The protocol included strengthening exercise with an intensity calculated by 1 Repetition maximum method technique11. Exercises were performed three days/ week (every alternate day), and the time required for single-day training is the time needed to complete 3 sets of 10 repetitions of each major muscle group.

High-Intensity Interval Training The HIIT protocol consisted of 10 s of the sprint, working at 85%- 90% of HRmax and 10 s of the recovery phase, during which participants cycled as slowly as possible for a total duration of 20 minutes. Participants were instructed when to start and stop in each phase. The duration of the exercise session was calculated for each participant individually.

1/2- High-Intensity Interval Training Participants in the 1/2-HIIT group followed the same protocol as the HIIT group, but only for the duration of 10 minutes working at 85%- 90% of HRmax of 12 s of sprint and 8 s of recovery phase.

Cool Down The cool-down session lasted for 5-10 minutes. During the period, full-body stretches were performed with low-intensity, long-hold stretching.

Exercise Termination Criteria

The exercise session was prematurely terminated on the occurrence of one of the following:

* Modified Borg dyspnea scale (RPP) at level 8 or above.
* Decrease in oxygen saturation<90%.
* Any complaints of chest pain, leg cramps, palpitation or tiredness by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Class I obese population BMI ≥25.0 -30.0
* Young adults aged 20-40 years
* Diagnosed patients with DM and dyslipidemia.

Exclusion Criteria:

-Patients diagnosed with pre-existing heart conditions, major illness (acute or chronic), beta-blockers, pregnant or lactating women, and smokers, including any that would limit the ability to perform the necessary exercises, will be excluded from the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Thyroid Stimulating Hormone | 16 weeks
  The levels of TSH were measured using blood sample (Biodata Diagnostic brand RIA kit)12. The samples were taken twice once before the start of the training protocol and second after the completion of 16 weeks of training. The difference in the values between the groups was used to evaluate the impact of exercises thyroid hormone levels in the body.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No